CLINICAL TRIAL: NCT07361198
Title: Percutaneous Transcatheter Genicular Embolization in Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENIEMB
Record Dates: First submitted 2025-12-30; First posted 2026-01-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritic Knee Pain; Osteo Arthritis of the Knee; Osteoarthitis
Keywords: genicular artery embolisation; osteoarthritis; MSK embolisation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with genicular artery embolisation (Experimental)
  Interventions: Procedure: genicular artery embolisation

INTERVENTIONS:
Procedure: genicular artery embolisation — The procedure will be performed in the angiography room under local anesthesia. After puncturing the common femoral artery, a microcatheter will be inserted into the arterial branches supplying the knee joint and DSA will be performed. The target lesions have a typical "blush" appearance representing pathological neovascularization. Embolization will be performed by applying a suspension of Imipenem/Cilastatin dissolved in saline with a contrast agent until flow in the target branch is stopped.

SUMMARY:
This clinical study investigates a minimally invasive treatment called percutaneous transcatheter embolization of knee arteries for patients with chronic knee pain caused by advanced knee osteoarthritis or persistent pain after total knee replacement. Osteoarthritis of the knee is a common degenerative condition that can lead to long-term pain, reduced mobility, and decreased quality of life, and some patients do not achieve sufficient relief with standard treatments.

The study is based on the hypothesis that targeted embolization of small arteries supplying the inflamed tissues of the knee can safely reduce abnormal blood flow associated with inflammation, leading to pain relief and improved knee function. During the procedure, a thin catheter is guided through the blood vessels to the affected area of the knee, where a temporary embolic agent is administered to reduce pathological blood supply.

The aim of the study is to evaluate the safety and effectiveness of this procedure by assessing changes in pain intensity, knee function, and quality of life over a follow-up period of up to 24 months. The results of this study may help determine whether this minimally invasive approach can offer a new treatment option for patients who have limited alternatives for managing chronic knee pain

DETAILED DESCRIPTION:
This is a prospective, single-center, interventional pilot study designed to assess a catheter-based endovascular technique targeting pathological vascular changes associated with chronic knee pain. The intervention focuses on selective embolization of abnormal synovial and periarticular arterial branches identified by angiographic imaging as areas of increased perfusion related to inflammatory activity.

The procedure is performed in an angiography suite under local anesthesia. Vascular access is obtained via the common femoral artery, followed by selective catheterization of the arterial branches supplying the knee joint. Digital subtraction angiography is used to visualize hypervascular regions, typically seen as focal contrast enhancement ("blush"). These regions are considered targets for treatment. Embolization is carried out using a temporary embolic suspension administered through a microcatheter until adequate flow reduction in the target vessels is achieved, while preserving normal surrounding circulation.

Participants undergo standardized clinical and imaging assessments before the intervention and during scheduled follow-up visits over a two-year period. Follow-up evaluations are intended to capture longitudinal changes in clinical status and to monitor for any procedure-related adverse events. The study emphasizes procedural safety, technical feasibility, and post-interventional monitoring rather than comparison with alternative therapies.

Data collected during the study are analyzed using descriptive and paired statistical methods appropriate for an exploratory pilot design. The study is conducted in accordance with applicable ethical standards and regulatory requirements, with particular attention to patient safety, data protection, and transparency of reporting. The findings are expected to provide technical and clinical insights to inform future larger-scale studies and potential integration of this approach into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 80 years
* Clinical symptoms consistent with chronic knee pain
* Radiographically confirmed knee osteoarthritis of Kellgren-Lawrence grade II-IV or persistent knee pain following total knee arthroplasty
* Insufficient pain relief after standard conservative treatment (e.g., pharmacological therapy, physical therapy, or injections)
* Ability to understand the study procedures and provide written informed consent _ Willingness and ability to comply with the study procedures and follow-up schedule

Exclusion Criteria:

* Active local or systemic infection
* Known coagulation disorders or ongoing anticoagulation that cannot be safely interrupted
* Significant peripheral arterial disease affecting the lower limbs
* Known allergy or contraindication to iodinated contrast agents
* Severe renal impairment
* History of fibromyalgia or other generalized chronic pain syndromes that may confound pain assessment
* Pregnancy or breastfeeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
VAS (Visual Analog Scale) score | In 1st, 3rd, 6th, 12th and 24th month after the procedure.
  A VAS score for knee pain uses a 0-10 scale, where 0 means no pain, and 10 means the worst imaginable pain, helping quantify intensity, often categorized as mild (1-3), moderate (4-6), and severe (7-10) to assess pain levels or treatment effectiveness.
WOMAC ( Western Ontario and McMaster Universities Osteoarthritis Index) score | In 1st, 3rd, 6th, 12th and 24th month after the procedure.
  The total WOMAC score can range from 0 to 96, with a higher number indicating greater disease severity. The final number is calculated by adding up the points in three separate subscales that assess pain (0-20 points), stiffness (0-8 points), and knee joint function (0-68 points).
KOOS (Knee Injury and Osteoarthritis Outcome Score) score | In 1st, 3rd, 6th, 12th and 24th month after the procedure.
  The KOOS score is a patient-completed questionnaire assessing knee health and function across five areas: Pain, Symptoms (stiffness/swelling), Activities of Daily Living (ADL), Sport & Recreation, and Quality of Life (QoL). It uses a 0-100 scale (0=worst, 100=best) to track outcomes after knee injuries or arthritis, helping evaluate treatment effectiveness.

SECONDARY OUTCOMES:
Analgetics use | In 1st, 3rd, 6th, 12th and 24th month after the procedure.
  Amount of analgesic use in mg per day

CONTACTS AND LOCATIONS:
Locations (1):
- Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Yes. Individual participant data (IPD) that underlie the results reported in this study, after de-identification, will be shared. This includes clinical, procedural, and follow-up data necessary to reproduce the reported findings.
  Data will be shared in a secure manner, and access may require a data use agreement to ensure compliance with ethical standards and data protection regulations.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Individual participant data will be available for sharing beginning after publication of the primary study results and up to five (5) years following completion of the study.
Access Criteria: The data will be made available upon reasonable request to qualified researchers for scientifically sound proposals. Requests should include a brief description of the research objectives and a statistical analysis plan and will be reviewed by the principal investigator.

REFERENCES:
- [Background] Fleckenstein FN, Maleitzke T, Auer TA, Bolle P, Gebauer B, Winkler T, Collettini F. Genicular Artery Embolization for the Treatment of Symptomatic Knee Osteoarthritis. Radiology. 2025 Jul;316(1):e243648. doi: 10.1148/radiol.243648. No abstract available. PMID 40693933
- [Background] Bagla S, Piechowiak R, Sajan A, Orlando J, Hartman T, Isaacson A. Multicenter Randomized Sham Controlled Study of Genicular Artery Embolization for Knee Pain Secondary to Osteoarthritis. J Vasc Interv Radiol. 2022 Jan;33(1):2-10.e2. doi: 10.1016/j.jvir.2021.09.019. Epub 2021 Oct 2. PMID 34610422
- [Background] Okuno Y, Korchi AM, Shinjo T, Kato S. Transcatheter arterial embolization as a treatment for medial knee pain in patients with mild to moderate osteoarthritis. Cardiovasc Intervent Radiol. 2015 Apr;38(2):336-43. doi: 10.1007/s00270-014-0944-8. Epub 2014 Jul 4. PMID 24993956
- [Background] van Zadelhoff TA, Bos PK, Moelker A, Bierma-Zeinstra SMA, van der Heijden RA, Oei EHG. Genicular artery embolisation versus sham embolisation for symptomatic osteoarthritis of the knee: a randomised controlled trial. BMJ Open. 2024 Oct 1;14(10):e087047. doi: 10.1136/bmjopen-2024-087047. PMID 39353688

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT07361198/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT07361198/ICF_001.pdf